CLINICAL TRIAL: NCT06453148
Title: Prospective Clinical Registry of Heart Transplant Patients in Brazil
Brief Title: Brazilian Clinical Registry of Heart Transplantation
Acronym: HESTIA
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Other Study IDs: HESTIA REGISTRY
Record Dates: First submitted 2024-06-07; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Heart Transplant Failure and Rejection; Heart Transplant
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart Transplantation: Adults heart transplantation
  Interventions: Other: Non-interventions

INTERVENTIONS:
Other: Non-interventions — Usual care evaluations

SUMMARY:
Prospective cohort clinical study, registry-based, multicenter, national, with the consecutive inclusion of patients with a history of Heart Transplantation in Brazil. The clinical registry will involve the participation until 25 centers. Patients will be included up to 30 days after Heart Transplant surgery and will be followed for one year. Laboratory tests and clinical parameters wil be collected in two clinical visits (6mo and 12 mo). The outcomes evaluate will be the total hospitalizations and all-cause death. It is expected to include 730 patients with a 12-month follow-up from the day of the transplant surgery. The findings of the HESTIA Registry may guide the management of post-heart transplant patients, aiming at reducing morbidity and mortality within 12 months after heart transplant surgery.

DETAILED DESCRIPTION:
The study will include participants who have undergone heart transplantation at transplant centers across Brazil. Patients will be enrolled within the first 30 days after surgery and will be followed for one year.

The study will be participant-centered through clinical visits. There will be an admission visit and two additional visits: one at 6 months (V1) and another at 12 months (V2), which will be the closing visit

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old;
* Heart Transplantation within 30 days of both sexes;

Exclusion Criteria:

* Refusal to provide consent for the study;
* In the judgment of the local investigator, any difficulty accessing follow-up visits

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart transplant patients
Sampling Method: Probability Sample
Enrollment: 730 (Estimated)
Dates: Start 2024-08-25 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2027-08-25 (Estimated)

PRIMARY OUTCOMES:
Combined of total hospitalizations and all-causes deaths | 12 months
  Incidence of Hospitalization and death

SECONDARY OUTCOMES:
Individual components of the primary outcome; | 12 months
  Time to occurrence hospitalizations and death
Incidence of hospitalizations due to infections not related to the primary outcome; | 12 months
  Time to occurrence of infections
Vaccination rate; | 12 months
  All vaccines recommended rate
Incidence of organ rejection; | 12 months
  Time to occurrence of organ rejection
Cardiovascular mortality; Cardiovascular mortality | 12 months
  Time to first occurrence of cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bacal, PhD, Study Chair — Heart Transplantation Coordinator - Hospital Albert Einstein; Henrique A Fonseca, PhD, Principal Investigator — Head of Vaccines and Immunobiology Clinical Trial - ARO-EINSTEIN; Iascara Wozniak de Campos, PhD, Principal Investigator — Clinical Trialist - ARO - EINSTEIN; Luiz V Rizzo, PhD, Principal Investigator — Director - ARO - EINSTEIN
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No